CLINICAL TRIAL: NCT06396104
Title: The Effect of Mobilization With Movement Technique on the Stiffness of Cervical Muscles in Individuals With Mechanical Neck Pain: A Randomized Controlled Trial
Brief Title: Mobilization With Movement Technique on the Stiffness of Cervical Muscles in Individuals With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Collaborators: Istanbul Kent University (Other); Istanbul University - Cerrahpasa (Other); Istanbul Demiroglu Bilim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUC001
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-04

CONDITIONS: Neck Pain
Keywords: Neck Pain; Manual Therapy; Sham Treatment
MeSH Terms: conditions — Neck Pain | interventions — Movement

STUDY DESIGN:
Intervention Model Description: A Parallel, double blind, randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The physiotherapist who will apply the evaluation methods to be used in our study will be blind to the group distribution of the patients. Additionally, patients will be blind to the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with movement group (Experimental)
  Interventions: Other: Mobilisation with movement
- Sham group (Sham Comparator)
  Interventions: Other: Sham mobilisation

INTERVENTIONS:
Other: Mobilisation with movement — The physiotherapist places the medial edge of the thumb of one hand on the upper facet joint of the relevant segment, then applies superior-anterior slide to the facet joint by providing support with the thumb of the other hand. The 'gliding' movement is maintained while the patient actively performs the unilateral neck rotation movement and maintains it for a few seconds at the end of the movement. If joint movement is painful, attempts are made on the other facet joint of the same segment or on the spinous process. If this attempt does not immediately improve the patient's active joint motion, Mulligan Sustained Natural Apophyseal Glides (SNAG) will be applied to the upper part of the left zygapophysial joint, and in case of failure again, application will be made through the superior spinous process of the relevant segment. Painless joint movement will be applied in 6 repetitions and 3 sets.
  Arms: Mobilization with movement group
Other: Sham mobilisation — While the patients are sitting in a chair with a supported back, the spinal segment where pain is felt in neck joint movements will be determined. Without applying a sliding movement to this segment over the facet joint, only sensory input will be given and the patient will be asked to continue the active rotation movement and wait a few seconds at the end of the movement. The application will be completed as 6 repetitions and 3 sets.
  Arms: Sham group

SUMMARY:
Mobilisation with movement (Mulligan Sustained Natural Apophyseal Glides (SNAG)). method has been shown to have significant effects on pain, joint range of motion, and functionality in patients with neck pain. However, there is a lack of studies examining the effects of this technique on muscle stiffness associated with neck pain. Considering the immediate effects of a single session of lumbar SNAG application on lumbar muscle stiffness in patients with low back pain, it raises curiosity about the effects it would have on cervical spinal segments and surrounding muscles. The aim of this study is to investigate the immediate effects of Mulligan SNAG application on muscle stiffness, pain, and joint range of motion in patients with mechanical neck pain.

DETAILED DESCRIPTION:
This study is designed as a parallel double-blind randomized controlled trial. Patients will be divided into two groups: the Mobilization with Movement Group (MMG) and the Sham Group (SG). The MMG will receive cervical mobilization (SNAG) treatment. The SG, on the other hand, will receive active joint movements without the 'sliding' motion applied to the spinal segment. Prior to and immediately after the intervention, participants will undergo myometric evaluation of neck muscles, joint range of motion measurements, and pressure pain threshold measurements bilaterally, followed by assessment of the individual's pain and level of disability using questionnaires related to pain and pain-associated disability. A 2-minute break will be provided after the intervention before reassessment is conducted. Patients will not be followed up.

ELIGIBILITY:
Inclusion Criteria:

* Having widespread neck pain lasting more than 3 months
* Pain symptoms that increase with neck movements or palpation
* Volunteering to participate in the study

Exclusion Criteria:

* History of neck trauma
* Previous cervical surgery
* Cervical radiculopathy or myelopathy
* Fibromyalgia syndrome diagnosis
* Any physiotherapy intervention in the previous 12 months
* Sign of vertebrobasilar insufficiency
* Upper cervical spine ligament instability
* Those using steroids or muscle relaxants

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Muscle stiffness | Baseline and immediately after application.
  Muscle stiffness will be measured with MyotonPRO (Myoton SA, Tallinn, Estonia). A brief mechanical pulse is applied to the skin over the muscle and then quickly released. Stiffness (N/m) is a parameter related to the capacity to withstand an external force. The reliability of the device has been proven in healthy individuals.The measurement site will be marked on the skin with a pen. In all applications, MyotonPRO's probe will be placed perpendicular to the skin and 3 measurements will be recorded using the multi-scanning mode with 10 pulses 1 second apart, and the average of the 3 measurements will be used for analysis.
  Upper trapezius: Evaluation will be performed in prone position. Measurements are from the midpoint between the lateral edge of the acromion and the spinous process of C7.
  Sternocleidomastoid: Measurements will be made at the midpoint between the sternum and the mastoid protrusion, with individuals lying in a supine position with a soft pillow under the neck.

SECONDARY OUTCOMES:
Joint Range of Motion | Baseline and immediately after application.
  An dual digital inclinometer (ACUMAR Model 002; Lafayette Instrument Company, Lafayette, Indiana) will be used to measure cervical rotation. The device consists of two simple digital inclinometers connected to each other with the help of cables. Measured joint range of motions are displayed on the screen on the digital inclinometer.
Numeric Pain Rating Scale | Baseline and immediately after application.
  Pain intensity of patients with neck pain will be obtained with the Numerical Rating Scale, which is reported to be a reliable and valid scale in determining pain intensity in the literature. In the scale, 0 indicates no pain and 100 indicates unbearable pain.
Neck Disability Index | Baseline
  Neck Disability Index (NDI) was used to evaluate the level of disability due to neck pain, which is a reliable and valid scale to determine the disability level of patients with chronic mechanical neck pain. NDI consists of 10 sections: pain intensity, personal care, weight lifting, reading, headaches, concentration, working, driving, sleep, and recreation. The score in each section varies between 0 (no disability) and 5 (complete disability). The total score ranges from 0 (no disability) to 50 (complete disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kent University, Istanbul, Turkey (Türkiye)